CLINICAL TRIAL: NCT00808093
Title: Food Effect Study of GSK256073A in Healthy Subjects
Brief Title: Repeat Dose Food Effect Study of GSK256073F in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 106777
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Dyslipidaemias
Keywords: Food Effect; GSK256073F; TRIS Salt
MeSH Terms: interventions — 8-chloro-3-pentyl-1H-purine-2,6(3H,7H)-dione

ARMS (1):
- fixed sequence (Other): fixed sequence (14 days fasted followed by 14 days either high fat or standard meal
  Interventions: Drug: GSK256073

INTERVENTIONS:
Drug: GSK256073 — GSK256073 100 mg study drug

SUMMARY:
The purpose of this study is to compare the effects of fasting and fed conditions with repeat doses of GSK256073F in HVT subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female of non-childbearing potential between 18 and 55 years of age.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 3 days post-last dose.
* Body weight > 50 kg (110 pounds) and BMI within the range 19 - 31 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. An exception is acetaminophen which is allowed at doses of ≤ 2g/day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Systolic blood pressure < 100 mmHg or ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg at screening.
* History of significant cardiac arrhythmias
* Active peptic ulcer disease (PUD) and/or history of PUD within 1 year.
* Screening test positive for H. Pylori using the non-radioactive breath test.
* A serum uric acid concentration ≥ 8mg/dL
* History of gout and/or hyperuricemia
* History of Gilbert's syndrome
* A serum creatinine concentration above the normal reference range
* History of kidney stones
* PT and/or aPTT above the reference range
* History of recurrent indigestion, stomach upset or diarrhea
* Liver function tests (LFTs) or creatinine phosphokinase (CPK) 2X ULN
* Screening stool test positive for occult blood
* Screening peripheral blood smear with abnormal RBCs
* Reduced G6PD activity
* Serum haptoglobin outside the reference range at screening
* Total serum LDH > 1.25% above the ULN at screening
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening (between the normal reference range up to 200ng/mL).
* History of flushing (>1 episode annually)
* Fasting blood glucose ≥ 110 mg/dl and/or history of type I or type II DM
* History of intra-ocular pathology, including but not limited to retinitis, uveitis, retinal detachment and macular edema
* History of recurrent gum bleeding
* History of bleeding haemorrhoids

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05-12 (Actual); Primary Completion 2008-08-27 (Actual); Study Completion 2008-08-27 (Actual)

PRIMARY OUTCOMES:
1. AUC0-inf, Cmax, and Ctrough (Ct) under fasting conditions | throughout study
2. AUC0-inf, Cmax, and Ctrough (Ct) under fed conditions | throughout the study

SECONDARY OUTCOMES:
1. Safety and tolerability will be assessed by vital signs, ECGs, clinical laboratory data, spontaneous AE reporting, nursing/physician observation and assessment of flushing via a visual analog scale | throughout the study
2. Tmax, t½ (if data permits), Ae (amount excreted in the urine), CLr (renal clearance), Cmax, ss, and Cτ following repeat dose | throughout the study
3. Pharmacodynamic endpoints may include TC, NEFA, HDL, LDL, TG, ApoA1, ApoA2, ApoB, Lp(a), CETP, adiponectin, liposcience (particle sizing) or other markers of dyslipidemia on Days 1, 14, 21, and 28, as data permit. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States